CLINICAL TRIAL: NCT00375453
Title: Phase I, Open-label, Dose Escalation Study for Evaluation of Safety, Tolerability, Pharmacokinetics, and Tumor-suppressive Efficacy of SH U04722 in Patients With Solid Tumors
Brief Title: Dose Escalation Study of SH U04722 in Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91526; 310681
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Tumors
Keywords: Paclitaxel; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: SH U04722

INTERVENTIONS:
Drug: SH U04722

SUMMARY:
This study will evaluate the safety and tolerability of SH U04722 in patients with solid tumor cancers. In addition, this study will identify the recommended dose and administration schedule of SH U04722 for phase II development in Japanese cancer patients, evaluate the pharmacokinetic profile of SH U04722 and gather preliminary data on the effectiveness of SH U04722 in patients with solid tumors.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:-Refractory to conventional antineoplastic treatment or no standard therapy option available-ECOG Performance Status score of < 2-Agreement not to take vitamin E products such as Juvela (except for over-the-counter [OTC] and diet supplements). Exclusion Criteria:- Patients treated with other unapproved drugs/investigational drugs, chemotherapy, biological response modifiers, immunotherapy or endocrinotherapy within 4 weeks prior to entry in this study or nitrosoureas within 6 weeks before initial dosing of SH U04722 -Patients on concurrent therapy with warfarin or coumarin derivatives.-Patients who had radiation therapy within 2 weeks prior to entry into this study. -Patients with a history of serious hypersensitivity to taxanes.-Patients with current peripheral neuropathy (? Common Terminology Criteria for Adverse Events [CTCAE] Grade 2)

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The number of patients with dose limiting toxicity (DLT) observed between Days 1 and 21 after start of treatment (after first 3 weekly administrations of SH U04722 plus 7 days)

SECONDARY OUTCOMES:
The number of patients with DLT observed by the end of Week 8
dose intensity (whether or not 75% of the planned dose can be done) for 8 weeks after the first dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Japan (3):
  - Hidaka-shi, Saitama
  - Iruma-gun, Saitama
  - Koutou-ku, Tokyo